CLINICAL TRIAL: NCT02666287
Title: An Open Label, Six-period Cross-over, Single and Repeat Dose Study to Determine the Pharmacokinetics of Fluticasone Furoate and GSK961081 When Administered Alone, in Combination, or Concurrently Via the ELLIPTA
Brief Title: GSK961081 Alone and With Fluticasone Furoate (FF), Phase 1 (Ph1), Single Dose Regimen (SD), Repeat Dose Regimen (RD), Pharmacokinetic (PK) Study in Healthy Volunteer (HV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201958
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Fluticasone furoate; Chronic obstructive pulmonary disease; Batefenterol; Dry Powder Inhaler; Respiratory; Pharmacokinetics; Ellipta; Healthy Subjects
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Each subject will receive all the 9 treatment regimens in the following order: A,G/B/F/C,H/E/D,I with a washout period of 7 days between each treatment period administered via the ELLIPTA inhaler. Where Treatment A= BAT/FF 900/300 microgram (mcg) (3 inhalations of 300/100 mcg).
  Treatment B= BAT 900 mcg (3 inhalations of 300 mcg) concurrently with FF (lactose) 300 mcg (3 inhalations of 100 mcg) from separate inhalers.
  Treatment C= BAT 900 mcg (3 inhalations of 300 mcg). Treatment D= FF (lactose) 300 mcg (3 inhalations of 100 mcg). Treatment E= FF (magnesium stearate [MgSt]) 300 mcg (3 inhalations of 100 mcg). Treatment F= FF/VI 300/75 mcg (3 inhalations of 100 mcg/25 mcg). Treatment G= 7-day repeat doses: BAT/FF 300/100 mcg (1 inhalation). Treatment H= 7-day repeat doses: BAT 300 mcg (1 inhalation). Treatment I= 7-day repeat doses: FF (lactose) 100 mcg (1 inhalation).
  Interventions: Drug: BAT/FF; Drug: BAT; Drug: FF; Drug: FF (MgSt); Drug: FF/Vilanterol
- Sequence 2 (Experimental): Each subject will receive all the 9 treatment regimens in the following order: B/C,H/A,G/D,I/F/E with a washout period of 7 days between each treatment period.
  Interventions: Drug: BAT/FF; Drug: BAT; Drug: FF; Drug: FF (MgSt); Drug: FF/Vilanterol
- Sequence 3 (Experimental): Each subject will receive all the 9 treatment regimens in the following order: C,H/D,I/B/E/A,G/F with a washout period of 7 days between each treatment period.
  Interventions: Drug: BAT/FF; Drug: BAT; Drug: FF; Drug: FF (MgSt); Drug: FF/Vilanterol
- Sequence 4 (Experimental): Each subject will receive all the 9 treatment regimens in the following order: D,I/E/C,H/F/B/A,G with a washout period of 7 days between each treatment period.
  Interventions: Drug: BAT/FF; Drug: BAT; Drug: FF; Drug: FF (MgSt); Drug: FF/Vilanterol
- Sequence 5 (Experimental): Each subject will receive all the 9 treatment regimens in the following order: E/F/D,I/A,G/C,H/B with a washout period of 7 days between each treatment period.
  Interventions: Drug: BAT/FF; Drug: BAT; Drug: FF; Drug: FF (MgSt); Drug: FF/Vilanterol
- Sequence 6 (Experimental): Each subject will receive all the 9 treatment regimens in the following order: F/A,G/E/B/D,I/C,H with a washout period of 7 days between each treatment period.
  Interventions: Drug: BAT/FF; Drug: BAT; Drug: FF; Drug: FF (MgSt); Drug: FF/Vilanterol

INTERVENTIONS:
Drug: BAT/FF — BAT/FF is available in DPI form and will be administered via the ELLIPTA inhaler. Each first strip contains 300 mcg per blister of BAT blended with lactose and its physical appearance is dry white powder. Second strip contains 100 mcg per blister of FF blended with lactose and its physical appearance is dry white powder.
Drug: BAT — BAT is available in DPI form and will be administered via the ELLIPTA inhaler. Each first strip contains 300 mcg per blister of BAT blended with lactose appear as dry white powder. Second strip contains lactose which appear as a dry white powder.
Drug: FF — FF is available in DPI form and will be administered via the ELLIPTA inhaler. Each first strip contains 100 mcg per blister of FF blended with lactose appear as dry white powder and second strip contains lactose which appear as dry white powder.
Drug: FF (MgSt) — FF magnesium stearate is available in DPI form and will be administered via the ELLIPTA inhaler. Each first strip contains 100 mcg per blister of FF blended with lactose appear as dry white powder and second strip contains lactose with magnesium stearate which appear as dry white powder.
Drug: FF/Vilanterol — FF/Vilanterol is available in DPI form and will be administered via the ELLIPTA inhaler. Each first strip contains 25 mcg per blister of vilanterol blended with lactose and magnesium stearate appear as dry white powder and second strip contains 100 mcg per blister of FF blended with lactose which appear as dry white powder.

SUMMARY:
Batefenterol (BAT) is a novel bifunctional molecule that combines muscarinic antagonism and beta2-agonism in a single molecule and is in development for the treatment of chronic obstructive pulmonary disease (COPD). FF is a corticosteroid approved as the inhaled corticosteroid (ICS) component of a combination product, with vilanterol (VI), a long-acting beta2-agonist for COPD. In the current study FF will be investigated as an inhaled product in combination with BAT, for treatment of COPD.

This study is an open-label, six-way crossover, single and repeat dose study to evaluate the systemic pharmacokinetics, safety and tolerability of FF and BAT when administered via the ELLIPTA™ alone, in combination, or concurrently at 3 times the clinical dose, following a single dose, and at the proposed clinical dose, following repeat doses.

This study will consist of screening period, 6 treatment periods, and a follow-up visit. Each subject will have 3 periods in which they receive a single dose treatment regimen (3 inhalations on Day 1 of each single dose study period) and 3 periods in which they receive a single dose treatment regimen followed by a 7-day, once-daily, repeated dose. On Day 1 of those periods, subjects will receive their single dose as 3 inhalations. On Days 2-8, subjects will receive 1 inhalation per day for the repeated dose regimen. There will be a minimum of 7-day washout between each treatment periods. All subjects will receive 9 treatments and follow-up procedures will be done 7 14 days after the last dose.

Forty eight healthy subjects will be enrolled into the study, such that approximately 40 subjects complete dosing and PK assessments. The total duration of participation for each subject in this study will be up to 15 weeks. ELLIPTA is a registered trademark of the GlaxoSmithKline [GSK] group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 64 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body mass index (BMI) within the range 18.5-30.0 kilogram per meter square (kg/m^2) inclusive.
* Male or female:

Males: Male subjects with female partners of child bearing potential must use a condom from the time of first dose of study medication until follow-up, or have had a vasectomy with documentation of azoospermia.

Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: Pre-menopausal females with one of the following: documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, documented bilateral oophorectomy.

Post-menopausal defined as 12 months of spontaneous amenorrhea, with simultaneous follicle stimulating hormone (FSH) and oestradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) during the trial, and until follow-up. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form as described in this protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Mean QTC > 450 millisecond (msec). NOTES: The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine read or manually over-read.

The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.

For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used as specified in the reporting and analysis plan (RAP).

* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or 12-lead ECG.
* Pre-existing condition(s) interfering with normal gastrointestinal (GI) anatomy or motility, including constipation, malabsorption or other GI dysfunction which may interfere with the absorption, distribution, metabolism or elimination of the study drug. Subjects with a history of cholecystectomy must be excluded.
* At screening, a supine blood pressure (BP) that is persistently higher (the mean of triplicate measurements taken at least 2 min apart) than 140/90 millimetres of mercury (mmHg).
* At screening, a supine mean (triplicate measurements) heart rate (HR) outside the range 40-90 beats per minute (bpm).
* Subject is mentally or legally incapacitated.
* A history of respiratory disease in the last 10 years.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study medication, unless in the opinion of the investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >21 units for males and >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 milliliter [mL]) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking; current smoker; or ex-smokers who (1) gave up less than 6 months ago or (2) who have a history of more than 10 pack-years. Pack-years is equal to cigarettes per day multiplied to number of years smoked divided by 20.
* History of sensitivity to any of the study medications or their components (beta agonist, anti-muscarinic, corticosteroid medication, magnesium stearate, or lactose), or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicated the subject's participation.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening or within 3 months before the first dose of study treatment.
* A positive test for human immunodeficiency virus (HIV).
* A positive pre-study drug/alcohol screen.
* The subject has participated in a clinical trial and has received an investigational product (IP) within 3 months before their first dose in the current study.
* Exposure to more than four new chemical entities within 12 months before the subject's first dose.
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days before the first dose of study medication until the follow-up visit.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-06-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of FF in plasma on Day 7 of repeat dosing | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dosing on Day 7 of each repeat dose regimen
  The following PK parameter will be measured: AUC
Maximum observed plasma concentration (Cmax) of FF in plasma on Day 7 of repeat dosing | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dosing on Day 7 of each repeat dose regimen
  The following PK parameter will be measured: Cmax

SECONDARY OUTCOMES:
AUC of BAT in plasma on Day 7 of repeat dosing | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dosing on Day 7 of each repeat dose regimen
Cmax of BAT in plasma on Day 7 of repeat dosing | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dosing on Day 7 of each repeat dose regimen
AUC of FF in plasma on Day 1 of study period | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dosing on Day 1 of each treatment period
Cmax of FF in plasma on Day 1 of study period | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dosing on Day 1 of each treatment period
AUC of BAT in plasma on Day 1 of study period | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dosing on Day 1 of each treatment period
Cmax of BAT in plasma on Day 1 of study period | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dosing on Day 1 of each treatment period
Number of participants with adverse events (AEs) | Up to 15 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Safety as assessed by 12-lead Electrocardiogram (ECG) | Up to 15 weeks
  A single 12-lead ECG will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and corrected QT (QTc) intervals.
Safety as assessed by systolic and diastolic blood pressure measurements | Up to 15 weeks
  Three readings of systolic and diastolic pressure will be taken at screening and Day -1. Single measurements will be taken at all other specified timepoints
Safety as assessed by oral temperature measurements | Up to 15 weeks
  Oral temperature measurements will be recorded at pre-dose on dosing days
Safety as assessed by heart rate measurements | Up to 15 weeks
  Three readings of heart rate will be taken at screening and Day -1. Single measurements will be taken at all other timepoints
Safety as assessed by respiratory rate measurements | Up to 15 weeks
  Respiratory rate measurements will be recorded at pre-dose on dosing days
Composite of Haematology parameters as a measure of safety | Up to 15 weeks
  The following hematology parameters will be measured: Platelet Count, red blood cell (RBC) count, Hemoglobin, Hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), white blood cell (WBC) count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils
Composite of Clinical Chemistry parameters as a measure of safety | Up to 15 weeks
  The following clinical chemistry parameters will be measured: Urea, Creatinine, Glucose (fasting), Uric acid, Potassium, Sodium, Calcium, Chloride, Phosphate, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase, Gamma-glutamyl transferase (GGT), Cholesterol, Triglycerides, Total Bilirubin, Total Protein, Albumin, and Globulin.
Composite of Urinalysis parameters as a measure of safety | Up to 15 weeks
  The following urinalysis parameters will be measured by dip stick test: protein, blood, ketones, glucose, bilirubin, urobilinogen, leukocyte esterase, specific gravity, nitrites, power of hydrogen (pH). If urine dipstick is abnormal for leukocyte esterase, nitrites, blood or protein, microscopic examination will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Ambery C, Young G, Fuller T, Georgiou A, Ramsay D, Puri A, Daley-Yates P. Open-Label, Crossover Study to Determine the Pharmacokinetics of Fluticasone Furoate and Batefenterol When Administered Alone, in Combination, or Concurrently. Clin Pharmacol Drug Dev. 2019 Feb;8(2):188-197. doi: 10.1002/cpdd.603. Epub 2018 Aug 2. PMID 30070770
- See also: Results for study 201958 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201958?search=study&search_terms=201958#rs